CLINICAL TRIAL: NCT00233480
Title: A Double-blind Randomized, Placebo-Controlled, Single-Center Study to Assess the Impact of Statins on the Autonomic Nervous System and Cardiac Structure/Function in Non-Ischemic Heart Failure
Brief Title: Statin Therapy in Heart Failure: Potential Mechanisms of Benefit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Pfizer (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Tamara Horwich, Tamara Horwich, MD, MS, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCLA IRB #04-12-007-01; 1K23HL085097-01A1 (NIH)
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Results first posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure, Congestive
Keywords: Randomized Controlled Trial; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Sympathetic Nervous System; Ventricular Remodeling; Chemokines
MeSH Terms: conditions — Heart Failure; Ventricular Remodeling | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active treatment (Experimental): atorvastatin 10mg QD x 3 months
  Interventions: Drug: atorvastatin
- placebo (Placebo Comparator): matched placebo QD x 3 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: atorvastatin — atorvastatin 10mg PO QD
  Other Names: lipitor
  Arms: active treatment
Drug: placebo — matched placebo Qd x 3 months
  Arms: placebo

SUMMARY:
The goal of the investigators' study is to further understand the potentially beneficial effects of statin therapy in patients with heart failure. It is hypothesized that statins will 1) increase the heart's pumping ability 2) improve functioning of the sympathetic nervous system and 3) decrease immune activation in heart failure.

DETAILED DESCRIPTION:
Recent evidence suggests that HMG-Coenzyme A (statin) therapy may be associated with improved survival in both ischemic and non-ischemic heart failure (HF). Large, randomized outcome studies of statins in HF are currently underway, but these trials will not address underlying mechanisms. The aim of the study is to investigate statins' potentially beneficial mechanisms of action in HF, focusing on: 1) sympathetic nervous system activation and 2) myocardial remodeling, and 3) immune activation in heart failure.

Fifty patients with systolic HF of non-ischemic etiology from a single center will be randomized in a double-blinded fashion to 3 months of atorvastatin 10mg QD (25 subjects) vs matching placebo QD (25 subjects). The following exams will be performed at baseline (pre-treatment) and at end of study (post-treatment): sympathetic microneurography, echocardiography, and peripheral blood chemokine analysis. Sympathetic microneurography at the peroneal nerve will directly quantify changes in sympathetic nerve activity (bursts/minute). Echocardiography (with the addition of MRI in a subset of subjects without pacemakers or implantable defibrillators) will be used to track changes in cardiac structure and function; indices of remodeling will include measurement of left ventricular mass index, left ventricular volume indices, left ventricular ejection fraction, and subendocardial scar quantification (MRI only). Immune activation will be characterized by circulating cytokines and chemokines. Additionally, quantification of established cardiac biomarkers (cardiac troponin, B-type natriuretic peptide, and C-reactive Protein), Holter monitor/heart rate variability studies, and quality of life and global clinical assessment will be performed pre- and post- treatment.

Neither sympathetic microneurography nor MRI have been previously utilized to assess statins' effects in humans with HF. The impact of statin therapy on inflammatory chemokine activation in HF also has not been studied. The knowledge gained from our proposed investigations may serve as a basis for understanding how statin therapy has potential to improve clinical outcomes in HF, and may ultimately lead to new therapeutic strategies for HF.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old
* LVEF ≤ 35%, as documented by echocardiography, radionuclide ventriculography, gated SPECT, or contrast ventriculography within past 6 months
* Symptomatic HF (NYHA II-IV) or current NYHA I with history of symptomatic HF within the last year
* Stable doses of optimal HF medical therapy, unless documented contraindication.

Exclusion Criteria:

* Ischemic etiology of HF, defined as the presence of at least one of the following four criteria; angiographic evidence of > 50% lesion in 1 or more of the 3 major epicardial vessels; history of myocardial infarction; history of revascularization procedure; evidence of significant perfusion defect in the setting of ischemic symptoms.
* Clinical indication for statin treatment - coronary artery, cerebrovascular, or peripheral vascular disease
* Major cardiovascular event or surgical procedure within past 8 weeks
* LDL<70 mg/dL
* HF secondary to congenital heart disease or uncorrected valvular disease
* Treatment with statin within past 2 months
* Pregnancy
* Contraindication to statin: moderate liver disease, AST/ALT > 150 U/ L, known hypersensitivity
* Likely to receive heart transplant within 3 months
* Known peripheral or autonomic neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara B Horwich, MD, Principal Investigator — UCLA Division of Cardiology
Locations (1):
- Ahmanson-UCLA Cardiomyopathy Center, Los Angeles, California, United States

REFERENCES:
- [Background] Horwich TB, Middlekauff HR. Potential autonomic nervous system effects of statins in heart failure. Heart Fail Clin. 2008 Apr;4(2):163-70. doi: 10.1016/j.hfc.2008.01.004. PMID 18433696
- [Background] Horwich TB, MacLellan WR. Atorvastatin and statins in the treatment of heart failure. Expert Opin Pharmacother. 2007 Dec;8(17):3061-8. doi: 10.1517/14656566.8.17.3061. PMID 18001265
- [Result] PubMed ID 22041323
- [Derived] Horwich TB, Middlekauff HR, Maclellan WR, Fonarow GC. Statins do not significantly affect muscle sympathetic nerve activity in humans with nonischemic heart failure: a double-blind placebo-controlled trial. J Card Fail. 2011 Nov;17(11):879-86. doi: 10.1016/j.cardfail.2011.07.008. Epub 2011 Sep 3. PMID 22041323

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Treatment | Placebo
Started | 14 | 13
Completed | 14 | 12
Not Completed | 0 | 1
Not completed — Underwent status II heart transplant | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (14) | 49 (17) | 48 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 6 | 10 | 16
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: LVEF (Left Ventricular Ejection Fraction)
Description: Left ventricular ejection fraction was assessed by transthoracic echocardiography according to Simpson's rule (biplane method of disks).
Time Frame: baseline and three months
Measure: Mean (Standard Error); unit: percent ejection fraction
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 14 | 12
percent ejection fraction
  Baseline LVEF | 24 (6) | 28 (7)
  3 month LVEF | 25 (6) | 24 (7)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; p = 0.025, paired t test

2. Primary Outcome: Muscle Sympathetic Nerve Activity (by Sympathetic Microneurography)
Time Frame: Baseline and three months
Population: Eighteen subjects had baseline and final sympathetic microneurographic tracings that were technically adequate for analysis. Reasons for inadequate microneurographic tracing were: 1) inability of investigators to locate sympathetic nerve on baseline or final study; or 2) inability of patient to tolerate discomfort of the procedure.
Measure: Mean (Standard Error); unit: bursts per minute
Groups:
- Active Treatment: atorvastatin 10mg daily for three months
- Placebo: matched placebo daily for three months
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 9 | 9
bursts per minute
  Baseline | 43 (3) | 39 (3)
  Three months | 36 (5) | 38 (3)

3. Secondary Outcome: Left Ventricular End-diastolic Dimension (LVEDD)
Description: The end-diastolic dimension of the left ventricle (in mm) was measured with 2D echocardiography performed by experienced technicians using Acuson Sequoia Echocardiography System
Time Frame: Baseline and three months
Measure: Mean (Standard Error); unit: Millimeters (mm)
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 14 | 12
Millimeters (mm)
  Baseline LVEDD | 65 (12) | 28 (7)
  Three months LVEDD | 25 (6) | 24 (7)

4. Secondary Outcome: Cardiac Biomarker Level BNP
Description: B-type natriuretic peptide, measured pg/mL at baseline and post-treatment
Time Frame: Baseline, 3 months
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 14 | 12
pg/mL
  Baseline | 175 [36 to 472] | 66 [29 to 154]
  Three Months | 107 [34 to 173] | 67 [21 to 299]

5. Secondary Outcome: High-sensitivity C-reactive Protein (hsCRP) as a Cardiac Biomarker
Time Frame: Baseline, Three months
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 14 | 12
mg/L
  Baseline | 1.6 [0.6 to 4.4] | 1.9 [1.0 to 3.0]
  Three months | 1.9 [.05 to 5.7] | 3.4 [1.1 to 5.9]

6. Secondary Outcome: Cardiac Troponin I (cTnI)
Description: Participants with cTnI ≥0.04 ng/mL
Time Frame: Baseline, Three months
Measure: Number; unit: percent of participants
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 14 | 12
percent of participants
  Baseline | 8 | 21
  Three Months | 0 | 15

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Active Treatment | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes